CLINICAL TRIAL: NCT03858413
Title: Correlation of a-Klotho Levels With the Severity of Calcification in the Coronary Arteries and Aortic Valve in Patients With Chronic Kidney Disease
Brief Title: a-Klotho in Relation to Calcification in the Coronary Arteries and Aortic Valve in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Panagiotis Savvoulidis, Principal Investigator, Royal Brompton & Harefield NHS Foundation Trust
Other Study IDs: 16/23-6-2016
Record Dates: First submitted 2019-02-22; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Vascular Calcification; Chronic Kidney Diseases
MeSH Terms: conditions — Vascular Calcification; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic kidney disease stage V: No intervention
  Interventions: Diagnostic Test: No intervention
- Chronic kidney disease stage III: No intervention
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
To define the correlation of the levels of a-Klotho with the severity of vascular calcification in the coronary arteries and aortic valve.

DETAILED DESCRIPTION:
Vascular calcification is a well-defined risk factor for cardiovascular disease and a-Klotho has been suggested to be an implicating factor in the process of vascular calcification, particularly in patients with chronic kidney disease (CKD).

With this study the investigators will examine the possible correlation of the levels of secreted a-Klotho with the severity of vascular calcification in the coronary arteries and aortic valve in patients with CKD at different stages of CKD. More precisely, a-Klotho was measured in 30 patients with end-stage renal disease under intermittent regular hemodialysis and 30 outpatients with stable CKD stage III (estimated glomerular filtration rate between 30 and 59 mL/min/1.73^2).

Participants in both groups were eligible only if stable for at least the last 3 months pre-enrollment. Calcification will be calculated using the well-established Agatston score after submitting all patients to multi-slice computed tomography.

Continuous variables will be described as median (25th-75th percentile) and categorical variables as N (%). Variables will be compared between groups using the non-parametric Mann-Whitney U test for continuous and Fisher's exact test for categorical variables. Bivariate correlations of a-Klotho levels with clinical variables and calcification scores using the Spearman correlation coefficient will be examined. Identification of a-Klotho determinants, log-transformation of a-Klotho levels was done because of log-normal distribution and stepwise linear regression was used, with probability to remove the variable>0.1. Identification of determinants of coronary and aortic calcification was done via log-transformation of the corresponding calcium scores, (a value of 0 was assumed; log-transformed-1 for absent calcium) and, stepwise linear regression was used as above. Because of the small sample size, all regression estimates, and confidence intervals were calculated with re-sampling so that robust variable selection and stable estimates can be ensured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic kidney disease stage V under intermittent hemodialysis and, patients with stable chronic kidney disease stage III

Exclusion Criteria:

* Active cancer
* Inflammatory or granulomatous disease
* Primary hyperparathyroidism
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two different populations have been selected. First group with patients with chronic kidney disease under hemodialysis. Second group with patients with chronic kidney disease stage III stable for the last at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Agatston score in coronary arteries. | During enrollment.
  Calcification of coronary arteries will be measured with multi-slice CT and dedicated software to calculate Agatston score.
  Initially, Hounsfield units will be measured and transformed into Agatston score net numbers.
  A brief description of the method is provided below:
  Method of calculation:
  The calculation is based on the weighted density score given to the highest attenuation value (HU) multiplied by the area of the calcification speck.
  Density factor: 130-199 HU: 1; 200-299 HU: 2; 300-399 HU: 3; 400+ HU: 4. The score of every calcified speck is summed up to give the total calcium score.
Agatston score in aortic valve. | During enrollment.
  Calcification aortic valve will be measured with multi-slice CT and dedicated software to calculate Agatston score.
  Initially, Hounsfield units will be measured and transformed into Agatston score net numbers.
  A brief description of the method is provided below:
  Method of calculation:
  The calculation is based on the weighted density score given to the highest attenuation value (HU) multiplied by the area of the calcification speck.
  Density factor: 130-199 HU: 1; 200-299 HU: 2; 300-399 HU: 3; 400+ HU: 4. The score of every calcified speck is summed up to give the total calcium score.
Circulating a-Klotho. | During enrollment.
  Circulating a-Klotho levels will be measured in serum with the use of a commercially available ELISA kit. Concentration will be expressed in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Hadjimiltiades, Professor, Study Director — Head of Interventional Cardiology Department

IPD SHARING:
Plan to Share IPD: No
No plans made to make IPD available to other researchers

REFERENCES:
- [Background] Kuro-o M, Matsumura Y, Aizawa H, Kawaguchi H, Suga T, Utsugi T, Ohyama Y, Kurabayashi M, Kaname T, Kume E, Iwasaki H, Iida A, Shiraki-Iida T, Nishikawa S, Nagai R, Nabeshima YI. Mutation of the mouse klotho gene leads to a syndrome resembling ageing. Nature. 1997 Nov 6;390(6655):45-51. doi: 10.1038/36285. PMID 9363890
- [Background] Shiraki-Iida T, Aizawa H, Matsumura Y, Sekine S, Iida A, Anazawa H, Nagai R, Kuro-o M, Nabeshima Y. Structure of the mouse klotho gene and its two transcripts encoding membrane and secreted protein. FEBS Lett. 1998 Mar 6;424(1-2):6-10. doi: 10.1016/s0014-5793(98)00127-6. PMID 9537505
- [Background] Olejnik A, Franczak A, Krzywonos-Zawadzka A, Kaluzna-Oleksy M, Bil-Lula I. The Biological Role of Klotho Protein in the Development of Cardiovascular Diseases. Biomed Res Int. 2018 Dec 24;2018:5171945. doi: 10.1155/2018/5171945. eCollection 2018. PMID 30671457
- [Background] Henaut L, Chillon JM, Kamel S, Massy ZA. Updates on the Mechanisms and the Care of Cardiovascular Calcification in Chronic Kidney Disease. Semin Nephrol. 2018 May;38(3):233-250. doi: 10.1016/j.semnephrol.2018.02.004. PMID 29753400
- [Background] Mencke R, Hillebrands JL; NIGRAM consortium. The role of the anti-ageing protein Klotho in vascular physiology and pathophysiology. Ageing Res Rev. 2017 May;35:124-146. doi: 10.1016/j.arr.2016.09.001. Epub 2016 Sep 28. PMID 27693241
- [Background] Navarro-Garcia JA, Fernandez-Velasco M, Delgado C, Delgado JF, Kuro-O M, Ruilope LM, Ruiz-Hurtado G. PTH, vitamin D, and the FGF-23-klotho axis and heart: Going beyond the confines of nephrology. Eur J Clin Invest. 2018 Apr;48(4). doi: 10.1111/eci.12902. Epub 2018 Feb 21. PMID 29394451
- [Background] Kuro-O M. The FGF23 and Klotho system beyond mineral metabolism. Clin Exp Nephrol. 2017 Mar;21(Suppl 1):64-69. doi: 10.1007/s10157-016-1357-6. Epub 2016 Nov 12. PMID 27838783
- [Background] Back M, Aranyi T, Cancela ML, Carracedo M, Conceicao N, Leftheriotis G, Macrae V, Martin L, Nitschke Y, Pasch A, Quaglino D, Rutsch F, Shanahan C, Sorribas V, Szeri F, Valdivielso P, Vanakker O, Kempf H. Endogenous Calcification Inhibitors in the Prevention of Vascular Calcification: A Consensus Statement From the COST Action EuroSoftCalcNet. Front Cardiovasc Med. 2019 Jan 18;5:196. doi: 10.3389/fcvm.2018.00196. eCollection 2018. PMID 30713844
- [Background] Olauson H, Mencke R, Hillebrands JL, Larsson TE. Tissue expression and source of circulating alphaKlotho. Bone. 2017 Jul;100:19-35. doi: 10.1016/j.bone.2017.03.043. Epub 2017 Mar 18. PMID 28323144